CLINICAL TRIAL: NCT03336034
Title: Assessment of Responsiveness to Treatment of the Experience Sampling Method (ESM) in Irritable Bowel Syndrome (IBS) Using Linaclotide
Brief Title: Assessment of Responsiveness to Treatment by Experience Sampling Method
Status: Terminated | Type: Observational
Why Stopped: Slow inclusion rate.
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: METC 173007; NL60925.068.17 (Registry Identifier: Toetsingonline)
Record Dates: First submitted 2017-10-25; First posted 2017-11-08 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Constipation-predominant Irritable Bowel Syndrome
Keywords: IBS-C; Experience sampling method; Ecological momentary assessment; Abdominal pain; Constipation
MeSH Terms: conditions — Abdominal Pain; Constipation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IBS-C: Constipation-predominant irritable bowel syndrome

SUMMARY:
Reliable evaluation of symptoms and their improvement during treatment is crucial in both diagnosing and evaluating response to treatment in IBS. Currently used end-of-day evaluations are considered sub-optimal and the Experience Sampling Method (ESM) was proposed previously as a more accurate symptom assessment method. Aim of this study is to evaluate the responsiveness of the developed ESM-PROM in assessing changes in abdominal pain and stool frequency after linaclotide treatment of IBS-C patients.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the internal and external responsiveness of the ESM-PROM in examining changes in symptom scores between baseline and post-treatment. Secondary objectives are to identify differences in characteristics between responders and non-responders to linaclotide and to assess for side effects of linaclotide treatment, using the ESM-PROM. This is a prospective, observational, single-group, open-label study, initiated and performed in Maastricht University Medical Center (MUMC+). The study population will conclude 30 IBS-C subjects that are newly prescribed with linaclotide by their treating physician at the outpatient department of gastroenterology and hepatology in the Maastricht UMC+. Primary study outcomes are the weekly average of the mean and maximum abdominal pain scores per day on the ESM-PROM per period (i.e. baseline, after 4 weeks and after 12 weeks). The ESM-PROM is completed during 7 consecutive days at each period and therefore, the measurements start one week before linaclotide treatment (baseline) and end one week after finishing linaclotide treatment (after 12 weeks). Further endpoints are the change scores of abdominal pain between pre- and post-treatment, measured using the ESM-PROM. Additionally, the proportion of overall responders to linaclotide treatment after 4 and 12 weeks assessed using the conventional end-of-day diary will be used to evaluate external responsiveness. Further endpoints are symptom scores as reported using the ESM-PROM, concerning abdominal pain, bloating, abdominal fullness, fecal urgency, stool consistency, straining, CSBM frequency and SBM frequency. Secondary outcomes are other factors measured using the ESM-PROM, i.e. non-GI physical symptoms, psychological status at the moment of symptom assessment, contextual information regarding the moment of symptom assessment as well as information on food and substance intake.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years;
* A diagnosis of IBS-C according to Rome IV criteria:

Recurrent abdominal pain, on average, at least 1 day per week in the last 3 months, associated with 2 or more of the following criteria: 1) Relation to defecation; 2) Association with a change in stool frequency; 3) Association with a change in stool form (appearance). Criteria fulfilled for the last 3 months with symptom onset at least 6 months ago. Reported stool consistency over the last 3 months: At least 25% of bowel movements are hard and lumpy stools (BSFS 1 or 2) and less than 25% of bowel movements are watery stools (BSFS 6 or 7).

* Negative colonoscopy in the past 5 years prior to inclusion;
* Treatment in primary care unsuccessful for 12 months;
* Ability to understand, read and speak the Dutch language;
* Ability to understand how to utilize the MEASuRE app on a smartphone.

Exclusion Criteria:

* Appendectomy or cholecystectomy within 2 months or other abdominal surgeries within 6 months before entry into the study;
* A history of laxative abuse;
* Current use of drugs that could initiate constipation (e.g. narcotics);
* Use of any IBS-related drugs possibly causing constipation (e.g. tricyclic antidepressants) are a reason for exclusion, unless usage is on a stable dose for at least 30 days before inclusion and there is no plan to change the dose during the study period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients visiting the outpatient department of the Division of Gastroenterology and Hepatology in MUMC+, diagnosed with constipation predominant irritable bowel syndrome (Rome IV), and newly prescribed with linaclotide 290µg once daily are eligible for inclusion.
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Mean abdominal pain scores as measured by the ESM tool. | 14 weeks (i.e. once during one week before linaclotide treatment, once during one week during linaclotide treatment and once during one week after the 12 week treatment period).
  Weekly average of mean abdominal pain scores per day on the ESM-PROM per period (i.e. baseline, after 4 weeks and after 12 weeks). Mean scores per day will be calculated, followed by calculating the mean of those 7 scores.
Maximum abdominal pain scores as measured by the ESM tool. | 14 weeks (i.e. once during one week before linaclotide treatment, once during one week during linaclotide treatment and once during one week after the 12 week treatment period).
  Weekly average of the maximum abdominal pain scores per day on the ESM-PROM per period (i.e. baseline, after 4 weeks and after 12 weeks). Maximum scores per day will be determined, followed by calculating the mean of those 7 scores.

SECONDARY OUTCOMES:
Number of bowel movements. | 14 weeks (i.e. once during one week before linaclotide treatment, once during one week during linaclotide treatment and once during one week after the 12 week treatment period).
  Number of complete spontaneous bowel movements per week, as measured by the ESM tool.
Symptom scores for other symptoms than abdominal pain, as measured by the ESM tool. | 14 weeks (i.e. once during one week before linaclotide treatment, once during one week during linaclotide treatment and once during one week after the 12 week treatment period).
  Symptom scores for non-GI physical symptoms, psychological symptoms, contextual information and information on food and drug intake.

CONTACTS AND LOCATIONS:
Overall Officials: Ad AM Masclee, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided